CLINICAL TRIAL: NCT06829576
Title: Comparative Examination of Health-related Physical Fitness in Individuals With Diabetic Dyslipidemia With Diabetic Individuals Without Dyslipidemia.
Brief Title: Examining Health-related Physical Fitness in Individuals With Diabetic Dyslipidemia.
Status: Completed | Type: Observational
Sponsor: Istanbul Galata University (Other)
Collaborators: Biruni University (Other)
Responsible Party: Principal Investigator, Safak Yigit, PT, PhD(c), Istanbul Galata University
Other Study IDs: GalataUni
Record Dates: First submitted 2025-01-31; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Dyslipidemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
To compare health-related physical fitness parameters in Type 2DM patients with and without dyslipidemia.Cardiometabolic biomarkers glucose and lipid profile will be noted from medical records. Body composition, functional capacity will be assessed with a six-minute walk test, peripheral muscle strength with a dynamometer, and physical activity level with a pedometer.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Type 2 DM for at least 1 year,

  * Having an HbA1c value between 6.5-11%,
  * Being between the ages of 35-65,
  * Knowing how to read and write Turkish,
  * Having signed the informed consent form

Exclusion Criteria:

* Lack of cooperation

  * Patients with peripheral or central serious neurological disorders
  * Patients with uncontrolled hypertension and uncontrolled arrhythmia
  * Pregnant or lactating patients
  * Patients with diabetic ulcers or neuropathy
  * Chronic renal failure (eGFR<30 ml/min)
  * Chronic liver disease (ALT/AST<3X Upper limit of normal)
  * Patients with serious respiratory system disease
  * Patients with cardiac pacemakers
  * History of previous stroke or myocardial infarction
  * Presence of lower and upper extremity orthopedic problems that may prevent the application of clinical tests

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Followed up in the Diabetes Polyclinic, Department of Internal Medicine, Endocrinology and Metabolic Diseases, Istanbul University, Istanbul Faculty of Medicine
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 1 day
  M. Quadriceps muscle strength and hand grip strength measurement will be used to evaluate peripheral muscle strength. Hand-held dynamometer will be used to evaluate quadriceps muscle strength and hand grip strength.
Funcitonal capacity | 1 day
  Submaximal functional exercise capacity of the participants will be evaluated with the six-minute walk test.
Waist circumference | 1 day
  Waist circumference will be measured at belly level with the patient in an upright position during expiration, with both feet bearing equal weight.
Hip circumference | 1 day
  Hip circumference will be measured at the level of the greater femoral trochanter, with the patient in an upright position, with both feet bearing equal weight.
Body fat-muscle ratios | 1 day
  Body fat-muscle ratios;These measurements will be determined by bioelectrical impedance.

SECONDARY OUTCOMES:
Physical activity level (step count) | 1 week (seven days)
  Step Count Measurement: Daily step count will be monitored to determine the physical activity level of the participants.Step count will be assessed with a wearable activity monitor, a portable, easy-to-use tool that can measure objectively (pedometer). With its six-axis sensor, the device records the user's physical activity style information in its temporary memory throughout the duration of use. After one week of use, the data recorded with the wearable activity monitor will be taken.
Glucose profile | 1 day
  Glucose profile, including Hemoglobin A1c (HbA1c) was measured. Additionally, the glucose profile will be assessed after 12 hours of fasting using standard biochemical analysis.
Glucose profile | 1 day
  Glucose profile, including fasting blood glucose (FBG), was measured. Additionally, the glucose profile will be assessed after 12 hours of fasting using standard biochemical analysis.
Lipid profile | 1 day
  Lipid profile, including low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), triglycerides (TG), and total cholesterol, will be measured after 12 hours of fasting using standard biochemical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akinci, Assoc.Prof, Study Director — Biruni University; Safak Yigit, PhD(c), Principal Investigator — Istanbul Galata University
Locations (1):
- Istanbul Galata University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No